CLINICAL TRIAL: NCT05788757
Title: A Post-Market Domestic (US) and International Data Collection to Assess the Optetrak Knee System
Brief Title: Optetrak Knee System Post Market Clinical Follow-Up
Status: Active, not recruiting | Type: Observational
Sponsor: Exactech (Industry)
Responsible Party: Sponsor
Other Study IDs: CR05-007
Record Dates: First submitted 2023-03-09; First posted 2023-03-29 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Knee Arthroplasty, Total

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Enrolled Subjects: Patients recruited from the population undergoing knee arthroplasty as part of standard of care. Patients who meet all the inclusion criteria and none of the exclusion criteria should be presented with an opportunity to undergo the informed consent process.
  Interventions: Device: Optetrak Total Knee System

INTERVENTIONS:
Device: Optetrak Total Knee System — Total Knee Arthroplasty using Exactech's Optetrak branded components.

SUMMARY:
A Post-Market Domestic (US) and International Data Collection to Assess the Optetrak Knee System

DETAILED DESCRIPTION:
Patient outcomes data is important for assessing the post-market safety and effectiveness of orthopedic medical devices. The purpose of this study is to collect clinical and patient outcomes and survivorship data for patients who have received or will receive a Optetrak® knee prosthesis manufactured or distributed by Exactech Inc (Gainesville, Florida, USA).

ELIGIBILITY:
Inclusion Criteria:

* Patient is indicated for knee replacement, or has already undergone knee replacement, with a device manufactured or distributed by Exactech
* Patient is skeletally mature
* Patient meets the indications detailed in the applicable product package insert Patient is willing and able to review and sign an informed consent form, if necessary

Exclusion Criteria:

* Patient has a local or systemic infection
* Patient has a known sensitivity to one or more of the materials in the knee replacement system to be used
* Patient is pregnant
* Patient has a mental or physical condition that may invalidate evaluation of the data - ---
* Patient is a prisoner
* Surgery is contraindicated according to the applicable product package insert

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must qualify for surgery per indications and contraindications as well as meet all the inclusion criteria and none of the exclusion criteria. The decision to offer a patient enrollment in this study is left to the discretion of the surgeon.
Sampling Method: Non-Probability Sample
Enrollment: 4588 (Estimated)
Dates: Start 2011-06-01 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2034-06-01 (Estimated)

PRIMARY OUTCOMES:
Knee Society Score | Preoperative
  (KSS) - validated outcome score
Knee Society Score | 6 month postoperative
  (KSS) - validated outcome score
Knee Society Score | annually through study completion, maximum of 10-years
  (KSS) - validated outcome score
Hospital for Special Surgery Knee Score | Preoperative
  (HSS) - validated outcome score
Hospital for Special Surgery Knee Score | 6 month postoperative
  (HSS) - validated outcome score
Hospital for Special Surgery Knee Score | annually through study completion, maximum of 10-years
  (HSS) - validated outcome score
Oxford Knee Score | Preoperative
  (OKS) - validated outcome score
Oxford Knee Score | 6 month postoperative
  (OKS) - validated outcome score
Oxford Knee Score | annually through study completion, maximum of 10-years
  (OKS) - validated outcome score

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Fallon Clinic, Worcester, Massachusetts
  - Nevada Orthopaedic and Spine Center, Las Vegas, Nevada
  - Medical University South Carolina, Charleston, South Carolina